CLINICAL TRIAL: NCT03617029
Title: Preoperative Localization With Microcoil Placement or Contrast Injection for Deep-seated Pulmonary Nodule : A Prospective Randomized Trial
Brief Title: Localization for Deep Lung Nodules: Microcoil Versus Contrast Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107-032-F
Record Dates: First submitted 2018-07-12; First posted 2018-08-06 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Lung Cancer
Keywords: Deep-seated; Needle localization; CT-guided; Thoracoscopy; Fiducial marker
MeSH Terms: conditions — Lung Neoplasms | interventions — Ethiodized Oil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microcoil (Experimental): Needle localization for deep-seated lung nodules with microcoil placement
  Interventions: Device: Microcoil
- Contrast (Active Comparator): Needle localization for deep-seated lung nodules with contrast injection
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Device: Microcoil — Needle localization with microcoil
  Arms: Microcoil
Drug: Lipiodol — Needle localization with contrast injection
  Arms: Contrast

SUMMARY:
In recent years, the development of low-dose pulmonary computed tomography screening has led to the discovery of many small pulmonary nodules in the early stages.

Surgical resection is still the main treatment for those suspected malignant lesions. In the face of such small pulmonary nodules, accurate preoperative localization has become the key to successful resection, and the deep-seated nodules are the most challenging parts. Because the deep-seated nodules cannot be localized by surface dye injection, however, it is necessary to place a fiducial marker (such as a microcoil) or contrast medium injection in combination with intraoperative fluoroscopy to ensure adequate resection of the deep-seated nodules. . This study will be carried out at the Hsinchu Branch of National Taiwan University Hospital. It is expected that 60 patients with pulmonary nodules with a depth larger than 2 cm will be randomly assigned into two groups. One group will receive microcoil placement, and the other group will receive contrast medium injection. The primary goal of the study was to compare the localization duration of the two groups of patients, the total dose of radiation exposure during localization and the incidence of location-related complications, and the secondary goals were the results of the surgical procedure, including the surgical duration.

ELIGIBILITY:
Inclusion Criteria:

Deep lung lesions

Exclusion Criteria:

Emphysema COPD Previous ilpislateral surgery

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Procedure success rate | 1 day
  Procedure success is defined as marking (lipiodol or hook-wire) the GGO lesion within 1 cm without pleural leakage of lipiodol or dislodgement of the hook-wire. The procedure success rate is calculated as follows: procedure success rate (%) = (number of procedure success / number of total procedure) × 100.
Successful localization for surgery | 1 day
  Localization contribute to surgery

SECONDARY OUTCOMES:
Procedure-related complication rate | 1 day
  Incidence of complications during needle procedure, The procedure-related complication rate is calculated as follows: procedure-related complication rate (%) = (number of procedure-related complication / number of total procedure) × 100.
Duration of the localization procedure | 1 day
  From start of needle procedure to withdraw of the needle (minutes)
Duration of wedge resection | 1 day
  From start of surgery to completion of pulmonary wedge resection (minutes)
Surgical margin of wedge resection | 1 day
  Distance from pulmonary lesion to resection margin of the specimen

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Hsin-Chu Branch, Taipei, Hsin-Chu County, Taiwan